CLINICAL TRIAL: NCT03046342
Title: Epidemiology of Acute Gastroenteritis in the Pediatric Population in Qatar: Causes, Risk Factors, Burden of Disease, Sources and Preventable Measures
Brief Title: Gastroenteritis in Pediatric Population of Qatar
Acronym: GE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-00045
Record Dates: First submitted 2017-01-31; First posted 2017-02-08 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2023-02

CONDITIONS: Gastroenteritis
Keywords: Gastroenteritis, Polymerase chain reaction
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Molecular method (PCR) — Stool samples are being processed through molecular method (PCR) for children with GE.
  Epidemiology of acute Gastroenteritis in the pediatric population in Qatar

SUMMARY:
Comparison of clinical and laboratory diagnosis for cause of Gastroenteritis(GE) depending on the clinical manifestation.Identifying the sources of viral, bacterial and parasitic GE in Pediatric population of Qatar

DETAILED DESCRIPTION:
Processing of stool samples by molecular method (PCR) for children with GE including complete data collection. Patients are followed up for 14 days

ELIGIBILITY:
Inclusion Criteria:

* All acute gastroenteritis patients between 3 months to 14 years presenting to PEC centers with acute diarrhea+/- vomiting with or without fever

Exclusion Criteria:

1. Cases of vomiting +/- fever only without diarrhea
2. Suspicion of surgical abdomen
3. Bile stained vomitus
4. Mal-absorption diseases as cystic fibrosis, celiac disease or increased secretion as disaccharides deficiency
5. Cases of Inflammatory bowel disease
6. Antibiotic associated diarrhea
7. Patients with immune deficiency
8. Patients with chronic diarrhea (>2 weeks of diarrhea)
9. Patients receiving long term medication for any disease

Ages: 3 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All acute gastroenteritis patients between 3 months to 14 years presenting to PEC centers with acute diarrhea+/- vomiting with or without fever
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-03-10 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
sources of viral, bacterial and parasitic GE in the country | 4 years
  Prevalence of viral, bacterial and parasitic GE in children < 14 years of age in Qatar will be identified by molecular method sample processing

SECONDARY OUTCOMES:
seasonal variation of GE in qatar determination | 4 years
  seasonal variation of GE in qatar being determined by number of cases reported during each season
comparing the prevalence of viral GE in vaccinated children in Qatar (against rotavirus) and the other countries which implemented rotavirus vaccine | 4 years
  comparing the prevalence of viral GE in vaccinated children in Qatar (against rotavirus) and the other countries which implemented rotavirus vaccine by detection of source of GE in vaccinated children by molecular method.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad medical corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No